CLINICAL TRIAL: NCT02036073
Title: Effect of Erythropoietin on Preterm Brain Injury
Acronym: EPO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhengzhou Children's Hospital, China (Other)
Collaborators: Zhengzhou University (Other)
Responsible Party: Principal Investigator, Huiqing Sun, Associate Professor, Zhengzhou Children's Hospital, China
Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CZZ-EPO
Record Dates: First submitted 2013-12-10; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Premature Birth
Keywords: erythropoietin; preterm; brain injury; cerebral palsy; PVL
MeSH Terms: conditions — Premature Birth; Brain Injuries; Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EPO (Experimental): In EPO group, the EPO was given by 500IU/kg every other day intravenously for 2 weeks. Recombinant human erythropoietin was configured by the hospital pharmacy intravenous Center Configuration, melted configured with saline to 1ml/kg solution. For severe patients, they were started to treat with EPO when their vital signs, blood pressure were stable.
  Interventions: Drug: recombinant human erythropoietin

INTERVENTIONS:
Drug: recombinant human erythropoietin — rhEPO 500U/kg was injected within 24h after birth, subsequent injection was given each other day fro 2 weeks.
  Other Names: EPO

SUMMARY:
EPO has been safely used for prevent preterm anemia and recent studies have shown the neuroprotective effect. Our hypothesis is that EPO could prevent preterm brain injury. The aims of this study include: to investigate the safety and efficacy of EPO by using 500u/kg higher than the dose of anemia treatment (250u/kg); to evaluate the effect of EPO on neurodevelopment in preterm infants; to detect biological indicators and explore the neuroprotective mechanism of EPO.

DETAILED DESCRIPTION:
Periventricular leukomalacia (PVL) is one of the most common brain injuries that occur in preterm infants, which is related with the development of cerebral palsy. The current therapy is only supportive to maintain the live sign stable. There is no effective therapeutic strategy for preterm brain injury. Erythropoietin (EPO) has been shown to be protective against hypoxic-ischemic and inflammatory injuries in animal models of brain injury, and clinical trials of neonatal hypoxic ischemic brain injury. Furthermore, recombinant human Epo (rhEpo) has been widely used in preterm infants to prevent or treat the anemia of prematurity during the past decade. It has been considered to be safe and well tolerated in preterm infants. However, there is no conclusion yet if the EPO has the effect to prevent preterm brain injury. The purpose of the study was whether the rhEpo (500 U/kg) given to very preterm infants (gestation age < 32 weeks) within 24h after birth and subsequently each other day for2 week possesses neuroprotective properties. Very preterm infants with gestational age of < 32 weeks and admit to our NICU are eligible for enrollment. After informed consent is obtained, infants will be randomly assigned to either EPO group or vehicle group. The primary short-term outcome measures are brain injury (intraventricular hemorrhage (IVH) and periventricular leukomalacia (PVL)) and ROP. The long term outcomes are whether rhEpo in very preterm infants finally improves neurodevelopmental outcome at 18 months corrected age.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants admitted to the NICU with gestational age <32 weeks
* birth weight <1500g and less than 72hours of age

Exclusion Criteria:

* 1. Infants with genetic metabolic diseases

  2. Congenital abnormalities

  3. Pneumothorax

  4. Grade III-IV intracranial hemorrhage

Ages: 1 Day to 72 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 490 (Actual)
Dates: Start 2009-01; Primary Completion 2012-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Incidence of MDI<70 | At corrected age of 18 months

SECONDARY OUTCOMES:
Incidence of ROP | At the corrected age 42 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zhengzhou Children's Hospital, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Sun H, Song J, Kang W, Wang Y, Sun X, Zhou C, Xiong H, Xu F, Li M, Zhang X, Yu Z, Peng X, Li B, Xu Y, Xing S, Wang X, Zhu C. Effect of early prophylactic low-dose recombinant human erythropoietin on retinopathy of prematurity in very preterm infants. J Transl Med. 2020 Oct 19;18(1):397. doi: 10.1186/s12967-020-02562-y. PMID 33076939